CLINICAL TRIAL: NCT04952090
Title: Development of Consciousness Measure and Monitor Device Based on Quantitative Electroencephalography Analysis In Emergency Patient
Brief Title: Development of Consciousness Measure and Monitor Device Based on Electroencephalography
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: National Research Foundation of Korea (Other)
Responsible Party: Sponsor
Other Study IDs: SNUEMS_HUMAN_EEG
Record Dates: First submitted 2021-06-20; First posted 2021-07-07 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2023-04

CONDITIONS: Electroencephalography; Consciousness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to develop a consciousness measuring and monitoring device using a single-channel electroencephalogram (EEG).

DETAILED DESCRIPTION:
Study objectives:

1. To develop a single-channel EEG database of emergency department (ED) patients with altered mental status.
2. To analyze single-channel EEG recordings and extract significant parameters.
3. To develop a consciousness prediction model using single-channel EEG.

Study design: observational multicenter study in 6 tertiary hospital EDs in Korea (Seoul National University Hospital, Seoul Metropolitan Government Seoul National University Boramae Medical Center, Kyungpook National University Hospital, Chungbuk National University Hospital, Chonnam National University Hospital, Korea University Ansan Hospital).

The investigators will obtain single-channel EEG data of ED patients with altered consciousness and develop a prospective database of the data.

With the constructed database, a consciousness prediction model using single-channel EEG will be developed.

The prediction performance of the developed model using area under receiver operating characteristic curve (AUC) will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Adult ED patients with a decreased level of consciousness (verbal, pain, or unresponsive using the AVPU scale, and a GCS-E score of less than 4) who have stayed at the ED for less than 12 hours at the time of enrollment.

Exclusion Criteria:

* Patients with the difficulty of applying EEG due to head trauma or skull deformities.
* Patients for whom standard treatment may be significantly delayed by applying the EEG device.
* Patients with a guardian who do not agree to enroll in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with a decreased level of consciousness who have visited the study hospital EDs and have stayed at the ED for less than 12 hours at the time of enrollment will be included.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2020-07-28 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Consciousness level using the Glasgow Coma Scale (GCS) scale. | At the time of study completion (May 31, 2023, anticipated).
  The GCS score ranges from 15 to 3 points, with a higher score indicating an alert consciousness and a lower score indicating decreased consciousness.
  A binary outcome of GCS<=8 and GCS>8 will be used in this study.

SECONDARY OUTCOMES:
Consciousness level using the AVPU (Alert; Verbal; Pain; Unresponsive) scale. | At the time of study completion (May 31, 2023, anticipated).
  A multi-class outcome (A: alert, V: verbal, P: pain, U: unresponsive) will be used in this study.

CONTACTS AND LOCATIONS:
Overall Officials: Ki Hong Kim, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea